CLINICAL TRIAL: NCT00789776
Title: A Phase I/II Study Evaluating the Safety and Efficacy of Adding a Single Prophylactic Donor Lymphocyte Infusion (DLI) of Natural Killer Cells Early After Nonmyeloablative, HLA-Haploidentical Hematopoietic Cell Transplantation - A Multi Center Trial
Brief Title: Fludarabine Phosphate, Cyclophosphamide, Total-Body Irradiation, and Donor Bone Marrow Transplant Followed by Donor Natural Killer Cell Therapy, Mycophenolate Mofetil, and Tacrolimus in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Wayne D. Kuni and Joan E. Kuni Foundation (Other)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2230.00; NCI-2010-00106 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2230.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Aggressive Non-Hodgkin Lymphoma; Diffuse Large B-Cell Lymphoma; Previously Treated Myelodysplastic Syndrome; Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Indolent Adult Non-Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Plasma Cell Myeloma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hodgkin Lymphoma; Refractory Plasma Cell Myeloma; Refractory Small Lymphocytic Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Mantle-Cell; Multiple Myeloma; Hodgkin Disease; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (non-myeloablative transplant) (Experimental): CONDITIONING: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total-body irradiation on day -1.
  DONOR BONE MARROW TRANSPLANTATION: Patients undergo donor bone marrow transplantation on day 0.
  POST-TRANSPLANTATION IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3 and mycophenolate mofetil PO TID on days 4 to 40, followed by a taper until day 84 in the absence of GVHD. Patients also receive tacrolimus IV continuously or IV QD over 1-2 hours or PO BID on days 4 to 84, followed by a taper until day 180 in the absence of GVHD.
  NK CELL INFUSION: Patients undergo donor lymphocyte infusion of NK cells on day 7.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Biological: Natural Killer Cell Therapy; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo donor bone marrow transplantation
  Other Names: Allo BMT; Allogeneic BMT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Biological: Natural Killer Cell Therapy — Given IV
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo total-body irradiation
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase I/II trial studies the side effects and best dose of donor natural killer (NK) cell therapy and to see how well it works when given together with fludarabine phosphate, cyclophosphamide, total-body irradiation, donor bone marrow transplant, mycophenolate mofetil, and tacrolimus in treating patients with hematologic cancer. Giving chemotherapy, such as fludarabine phosphate and cyclophosphamide, and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving an infusion of the donor's T cells (donor lymphocyte infusion) may help the patient's immune system see any remaining cancer cells as not belonging in the patient's body and destroy them (called graft-versus-tumor effect). Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving mycophenolate mofetil and tacrolimus after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identification of the maximal feasible dose of NK cells that can be infused one week after nonmyeloablative, human leukocyte antigen (HLA)-haploidentical hematopoietic cell transplant (HCT). (Phase I)

SECONDARY OBJECTIVES:

Once the maximal feasible dose has been identified, accrual will be limited to the cohort containing this cell dose to determine:

I. Incidence of relapse. (Phase II)

II. Incidence of grades III-IV acute graft-versus-host disease (GVHD). (Phase II)

III. Incidence of non-relapse mortality. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of donor NK cell therapy followed by a phase II study.

CONDITIONING: Patients receive fludarabine intravenously (IV) over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total-body irradiation on day -1.

DONOR BONE MARROW TRANSPLANTATION: Patients undergo donor bone marrow transplantation on day 0.

POST-TRANSPLANTATION IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3 and mycophenolate mofetil orally (PO) thrice daily (TID) on days 4 to 40, followed by a taper until day 84 in the absence of GVHD. Patients also receive tacrolimus IV continuously or IV once daily (QD) over 1-2 hours or PO twice daily (BID) on days 4 to 84, followed by a taper until day 180 in the absence of GVHD.

DONOR NK CELL INFUSION: Patients undergo donor lymphocyte infusion of NK cells on day 7.

After completion of study treatment, patients are followed up at 6 months, 1 year, 1.5 years, and then every year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following hematologic malignancies will be permitted although other diagnoses can be considered if approved by Patient Care Conference (PCC) and the principal investigators:
* Aggressive non-Hodgkin lymphomas (NHL) and other histologies such as diffuse large B cell (DLBC) NHL - a) not eligible for autologous HCT, b) not eligible for high-dose HCT, c) after failed autologous HCT, or d) be part of a tandem auto-allo approach for high risk patients
* Mantle cell NHL must be beyond first complete response (CR)
* Low-grade NHL with < 6 month duration of CR between courses of conventional therapy
* Chronic lymphocytic leukemia (CLL) must have either

  * 1) Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing FLU (fludarabine phosphate) (or another nucleoside analog, e.g. 2-chlorodeoxyadenosine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog)
  * 2) Failed FLU- CY (cyclophosphamide)-rituximab (FCR) combination chemotherapy at any time point; or
  * 3) Have "17p deletion" cytogenetic abnormality and relapsed at any time point after any initial chemotherapy
* Hodgkin lymphoma - must have received and a) failed frontline therapy, b) not be eligible for autologous HCT, or c) or be part of a tandem auto-allo approach for high risk patients
* Multiple myeloma or plasma cell leukemia must have received more than one line of prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HCT is permitted
* Acute myeloid leukemia (AML) must have < 5% marrow blasts at the time of HCT
* Acute lymphocytic leukemia (ALL) must have < 5% marrow blasts at the time of HCT
* Chronic myeloid leukemia (CML) accepted if they are beyond chronic phase (CP)1 and if they have received previous myelosuppressive chemotherapy or HCT and have < 5% marrow blasts at time of transplant
* Myelodysplasia (MDS)/myeloproliferative syndrome (MPS) - (> intermediate 1 [int-1] per International Prognostic Scoring System [IPSS]) after > or = 1 prior cycle of induction chemotherapy; must have < 5% marrow blasts at time of transplant
* Waldenstrom's macroglobulinemia must have failed 2 courses of therapy
* Patients must be expected to have disease controlled for at least 60 days after HCT
* Patients for whom HLA-matched unrelated donor search could not be initiated or completed due to insurance reasons, concerns of rapidly progressive disease, and/or discretion of attending physician are eligible for this protocol
* DONOR: Related, HLA-haploidentical donors who are identical for one HLA haplotype and mismatched for any number of HLA-A, -B, -C, DRB1 or DQB1 loci of the unshared haplotype
* DONOR: Marrow will be the only allowed hematopoietic stem cell source
* DONOR: Haploidentical donor selection will be based on standard institutional criteria, otherwise no specific prioritization will be made amongst the suitable available donors; donors will not be selected based on killer cell immunoglobulin-like receptor (KIR) status

Exclusion Criteria:

* Patients with available HLA-matched related donors
* Patients eligible for a curative autologous HCT
* Significant organ dysfunction that would prevent compliance with conditioning, GVHD prophylaxis, or would severely limit the probability of survival:

  * 1) Symptomatic coronary artery disease or ejection fraction < 35% or other cardiac failure requiring therapy (or, if unable to obtain ejection fraction, shortening fraction of < 26%); if shortening fraction is < 26% a cardiology consult is required with the principal investigator (PI) having final approval of eligibility
  * 2) Diffusion capacity of the lung for carbon monoxide (DLCO) < 40% total lung capacity (TLC) < 40%, forced expiratory volume in one second (FEV1) < 40% and/or receiving supplementary continuous oxygen; the Fred Hutchinson Cancer Research Center (FHCRC) study PI must approve enrollment of all patients with pulmonary nodules
  * 3) Liver function abnormalities: patient with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; the patient will be excluded if he/she is found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* Human immunodeficiency virus (HIV) seropositive patients
* Patients with poorly controlled hypertension despite multiple antihypertensive medications
* Fertile females who are unwilling to use contraceptive techniques during and for the twelve months following treatment, as well as females who are pregnant or actively breast feeding
* Fertile males who are unwilling to use contraceptive techniques during and for the twelve months following treatment
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers) or those with non-hematologic malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within five years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Active infectious disease concerns
* Karnofsky performance score < 60 Lansky performance score < 60
* Life expectancy severely limited by diseases other than malignancy
* Patients with a diagnosis of chronic myelomonocytic leukemia (CMML)
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Patients with AML, MDS, ALL, or CML must not have presence of circulating leukemic blasts detected by standard pathology
* Patients with aggressive lymphomas (such as DLBC) must not have bulky, rapidly progressive disease immediately prior to HCT
* Patients who have received a prior allogeneic HCT must have no active GVHD requiring immunosuppressive therapy for at least 21 days prior to start of conditioning
* DONOR: Children less than 12 years of age.
* DONOR: Children greater than or equal to 12 years of age who have not provided informed assent in the presence of a parent and an attending physician who is not a member of the recipient's care team
* DONOR: Children greater than or equal to 12 years of age who have inadequate peripheral vein access to safely undergo apheresis
* DONOR: Donors unable or unwilling to undergo marrow harvest for the initial HCT, storage of autologous blood prior to marrow harvest or apheresis one week after marrow harvest
* DONOR: Donors who are not expected to meet the minimum target dose of marrow cells (1 x 10^8 nucleated cells/kg recipient ideal body weight [IBW]) for the initial HCT; the average nucleated cell content of harvested marrow is 22 x 10^6 nucleated cells/mL or 220 x 10^8 nucleated cells/Liter
* DONOR: HIV-positive donors
* DONOR: Donors who are cross-match positive with recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-10-13 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose 1 (2.5 x 10^6/kg NK Cells): CONDITIONING: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total-body irradiation on day -1.
  DONOR BONE MARROW TRANSPLANTATION: Patients undergo donor bone marrow transplantation on day 0.
  POST-TRANSPLANTATION IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3 and mycophenolate mofetil PO TID on days 4 - 40, followed by a taper until day 84 in the absence of GVHD. Patients also receive tacrolimus IV continuously or IV QD over 1-2 hours or PO BID on days 4 - 84, followed by a taper until day 180 in the absence of GVHD.
  NK CELL INFUSION: Patients undergo donor lymphocyte infusion of 2.5 x 10^6/kg NK cells on day 7.
  Allogeneic Bone Marrow Transplantation: Undergo donor bone marrow transplantation
  Laboratory Biomarker Analysis: Correlative studies
- Dose 2 (5.0 x 10^6/kg NK Cells): CONDITIONING: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total-body irradiation on day -1.
  DONOR BONE MARROW TRANSPLANTATION: Patients undergo donor bone marrow transplantation on day 0.
  POST-TRANSPLANTATION IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3 and mycophenolate mofetil PO TID on days 4 - 40, followed by a taper until day 84 in the absence of GVHD. Patients also receive tacrolimus IV continuously or IV QD over 1-2 hours or PO BID on days 4 - 84, followed by a taper until day 180 in the absence of GVHD.
  NK CELL INFUSION: Patients undergo donor lymphocyte infusion of 5.0 x 10^6/kg NK cells on day 7.
  Allogeneic Bone Marrow Transplantation: Undergo donor bone marrow transplantation
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Started | 5 | 36
Completed | 5 | 35
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject aborted transplant after conditioning due to donor ineligibility. This subject was counted towards accrual but not evaluated with respect to outcome measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells) | Total
Number analyzed (Participants) | 5 | 36 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 10 | 11
  Between 18 and 65 years | 4 | 23 | 27
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Full Range); unit: years] | 22.2 [14.5 to 43.7] | 55.65 [8.1 to 75.2] | 47.6 [8.1 to 75.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 3 | 25 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 4 | 31 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 6 | 6
  White | 4 | 28 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 36 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Defined as having at least one of the following adverse events, independent of the attribution to the Natural Killer cell infusion: grade IV infusional toxicity (based on the Adapted Common Toxicity Criteria); grade IV regimen-related toxicity (based on Adapted Common Toxicity Criteria); grade IV acute Graft-Versus-Host Disease; non-relapse mortality.
Time Frame: Day 35 (28 days after NK cell infusion)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Relapsed Disease
Description: CML New cytogenetic abnormality and/or development of accelerated phase or blast crisis. The criteria for accelerated phase will be defined as unexplained fever greater than 38.3°C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, marrow blasts and promyelocytes >20%.
  AML, ALL >5% marrow blasts by morphologic or flow cytometric, or appearance of extramedullary disease.
  CLL ≥1 of: Physical exam/Imaging studies (nodes, liver, and/or spleen) ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ treatment; or definite increase in the size or number of plasmacytomas or lytic bone lesions.
Time Frame: At 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 1 | 10

3. Primary Outcome: Number of Participants With Grades III-IV Acute GVHD
Description: Number of patients who developed acute GVHD post-transplant. aGVHD Stages
  Skin:
  a maculopapular eruption involving < 25% BSA a maculopapular eruption involving 25 - 50% BSA generalized erythroderma generalized erythroderma with bullous formation and often with desquamation
  Liver:
  bilirubin 2.0 - 3.0 mg/100 mL bilirubin 3 - 5.9 mg/100 mL bilirubin 6 - 14.9 mg/100 mL bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: Day 100
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 1 | 0

4. Primary Outcome: Number of Non-relapse Participant Mortalities
Description: Defined as death in any patient for whom there has not been a diagnosis of relapse or disease progression.
Time Frame: Day 200
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 0 | 0

5. Primary Outcome: Number of Participants Who Experienced Graft Failure
Description: Graft failure is defined as grade IV thrombocytopenia and neutropenia after Day +21 that lasts >2 weeks and is refractory to growth factor support.
Time Frame: Day 100
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 0 | 4

6. Secondary Outcome: Number of Subjects Surviving Post-transplant.
Description: Number of subjects surviving post-transplant.
Time Frame: Up to 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 5 | 25

7. Secondary Outcome: Number of Participants Who Experienced Chronic Extensive GVHD
Description: Number of patients who developed chronic extensive GVHD post-transplant. The diagnosis of chronic GVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Time Frame: Up to 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
Number analyzed (Participants) | 5 | 35
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200; All-Cause Mortality: Conditioning through 1 Year.
Groups:
- Dose 1 (2.5 x 10^6/kg NK Cells); Dose 2 (5.0 x 10^6/kg NK Cells): CONDITIONING: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1 hour on days -6 and -5. Patients undergo total-body irradiation on day -1.
  DONOR BONE MARROW TRANSPLANTATION: Patients undergo donor bone marrow transplantation on day 0.
  POST-TRANSPLANTATION IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on day 3 and mycophenolate mofetil PO TID on days 4 - 40, followed by a taper until day 84 in the absence of GVHD. Patients also receive tacrolimus IV continuously or IV QD over 1-2 hours or PO BID on days 4 - 84, followed by a taper until day 180 in the absence of GVHD.
  NK CELL INFUSION: Patients undergo donor lymphocyte infusion of NK cells on day 7.
  Allogeneic Bone Marrow Transplantation: Undergo donor bone marrow transplantation
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Natural Killer Cell
Arm/Group | Dose 1 (2.5 x 10^6/kg NK Cells) | Dose 2 (5.0 x 10^6/kg NK Cells)
All-Cause Mortality (participants affected / at risk) | 0/5 | 10/35
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/35
Other Adverse Events (participants affected / at risk) | 4/5 | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (2.5 x 10^6/kg NK Cells) (N=5) | Dose 2 (5.0 x 10^6/kg NK Cells) (N=35)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (2.5 x 10^6/kg NK Cells) (N=5) | Dose 2 (5.0 x 10^6/kg NK Cells) (N=35)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (7)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (E. Coli & Klebsiella) (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Multiple) (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (viral/atypical bacterial infection vs. BOOP differenti (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Focal thrombotic microangiopathy found on renal bx) (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT00789776/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT00789776/Prot_SAP_001.pdf